CLINICAL TRIAL: NCT04094922
Title: PTSD Coach Sweden: Evaluating a Self-help Mobile App for Posttraumatic Stress in a Community Sample
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UU_neuro_kckp_PTSDcoach
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Posttraumatic Stress
Keywords: Posttraumatic Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Free access to the Swedish PTSD Coach smartphone app for three months.
  Interventions: Behavioral: Swedish PTSD Coach smartphone app
- Waitlist (No Intervention): Delayed access to the Swedish PTSD Coach smartphone app. Access is given after post-intervention data collection at three months.

INTERVENTIONS:
Behavioral: Swedish PTSD Coach smartphone app — Self-help smartphone app targeted towards posttraumatic stress that includes psychoeducation, rating/monitoring of distress, lists of support and treatment resources, and strategies for coping with distress.
  Arms: Intervention

SUMMARY:
Individuals who experience potentially traumatic events might develop long-lasting mental health problems. Limitations to health care resources, particularly in the context of mass disasters, indicate that self-help interventions could serve as important complementary offers to people in need.

The aim of this study is to evaluate whether the Swedish version of the Swedish version of the PTSD Coach self-help smartphone application can reduce levels of posttraumatic stress and related difficulties. The study is a randomized controlled trial in which participants' levels of posttraumatic stress and related difficulties after three months use of PTSD Coach will be compared to a waitlist condition. Additionally, in order to better understand the interplay between app use and health status, participants in both groups will receive text messages in which they are asked to respond to a small number of very brief questions about specific behaviors and current health status for three weeks during the intervention period.

DETAILED DESCRIPTION:
A majority of humans experience a potentially traumatic event during their lifetime, and many experience more than one. These events are of overwhelming emotional nature and have the capacity to evoke intensive distress. For many people, the distress dissipates either spontaneously or with the help from professional supports over the course of a couple of weeks. However, a substantial minority of people go on to develop significant levels of posttraumatic stress.

Chronic posttraumatic stress is often experienced together with clinical levels of other forms of psychopathology such as depression or anxiety disorders and the chronic condition can become debilitating over many years. There are effective interventions, however, they are as of yet difficult to access.

An uncontrolled pilot study of the Swedish PTSD Coach smartphone app indicated favorable outcomes and feasibility of the intervention (Cernvall, Sveen, Johannesson, & Arnberg, 2018). The app includes four modules: psychoeducation, rating and monitoring of distress, information about help and support, and strategies to cope with distress. The app is designed to be used with or without internet connection and uses little space on the smartphone.

This study will investigate whether the Swedish version of the PTSD Coach self-help smartphone application is beneficial for people who experience elevated levels of posttraumatic stress after a potentially traumatic event. The study is a randomized controlled trial with two conditions. In the intervention condition, participants are allowed free use of the PTSD Coach smartphone app. The control group is a waitlist condition. The intervention will take place during three months and is powered to detect a between-group effect size at the post-intervention assessment of d=0.5.

This study will also use an intensive longitudinal data collection method within the intervention period in order to better understand the interplay between app use and health status. Participants in both groups will receive text messages in which they are asked to respond to six very brief questions about specific behaviors and current health status for three weeks during the intervention period.

After the intervention period, participants across groups will be compared on a number of outcome variables related to posttraumatic stress, other mental health issues, daily function, and measures on healthcare consumption. The participants in the waitlist group will then be given access to the PTSD Coach app and both groups will be followed for two additional assessments after six and nine months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Adequate Swedish language comprehension
* Experienced a potentially traumatic event according to DSM-5 PTSD Criterion A during the past 2 years
* At least mild forms of posttraumatic stress, i.e., PCL-5 total score ≥ 10
* Access to smartphone able to run PTSD Coach app

Exclusion Criteria:

* Positive screening for bipolar disorder, psychotic disorder, ongoing substance disorder, or severe suicidality according to Mini International Neuropsychiatric Interview version 7.0.0
* current or planned psychological treatment within next three months
* current use of medication that may influence psychological treatment
* change in medication in the past months or planned changes within next three months
* ongoing potential traumatic context (e.g., ongoing domestic violence)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | 3 months (post)
  Self-report questionnaire for posttraumatic stress

SECONDARY OUTCOMES:
PTSD Checklist for DSM-5 | 6 months (3 months after intervention end)
  Self-report questionnaire for posttraumatic stress
PTSD Checklist for DSM-5 | 9 months (6 months after intervention end)
  Self-report questionnaire for posttraumatic stress
Patient Health Questionnaire (PHQ-9) | 3 months (post intervention)
  Self-report questionnaire for depressive symptoms
PHQ-9 | 6 months (3 months after intervention end)
  Self-report questionnaire for depressive symptoms
PHQ-9 | 9 months (6 months after intervention end)
  Self-report questionnaire for depressive symptoms
WHO Disability Assessment Schedule 2.0 (WHODAS) | 3 months (post intervention)
  Self-report questionnaire for functional disability, 12-item version
WHODAS | 6 months (3 months after intervention end)
  Self-report questionnaire for functional disability, 12-item version
WHODAS | 9 months (6 months after intervention end)
  Self-report questionnaire for functional disability, 12-item version
Trimbos Questionnaire for Costs (TiC-P) | 3 months (post intervention)
  Self-report questionnaire for healthcare use and productivity loss
TiC-P | 6 months (3 months after intervention end)
  Self-report questionnaire for healthcare use and productivity loss
TiC-P | 9 months (6 months after intervention end)
  Self-report questionnaire for healthcare use and productivity loss
Patient Health Questionnaire for physical symptoms (PHQ-15) | 3 months (post intervention)
  Self-report questionnaire for physical symptoms
PHQ-15 | 6 months (3 months after intervention end)
  Self-report questionnaire for physical symptoms
PHQ-15 | 9 months (6 months after intervention end)
  Self-report questionnaire for physical symptoms

OTHER OUTCOMES:
PTSD Coach Survey | 3 months (post intervention for intervention group); 6 months (post intervention for waitlist group)
  Self-report questionnaire to assess user satisfaction and perceived helpfulness of the app
Negative Effects Questionnaire (NEQ) | 3 months (post intervention for intervention group); 6 months (post intervention for waitlist group)
  Self-report questionnaire for negative effects related to the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Arnberg, PhD, Principal Investigator — Uppsala University
Locations (1):
- National Centre for Disaster Psychiatry, Department of Neuroscience, Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Cernvall M, Sveen J, Bergh Johannesson K, Arnberg F. A pilot study of user satisfaction and perceived helpfulness of the Swedish version of the mobile app PTSD Coach. Eur J Psychotraumatol. 2018 May 17;9(Suppl 1):1472990. doi: 10.1080/20008198.2018.1472990. eCollection 2018. PMID 29805783
- [Derived] Siverskog J, Andersson J, Hensler I, Gronqvist E, Arnberg FK. Cost-Effectiveness of App-Guided Self-Management for Posttraumatic Stress: Trial-Based Economic Evaluation. J Med Internet Res. 2025 Sep 18;27:e69426. doi: 10.2196/69426. PMID 40966669
- [Derived] Hensler I, Sveen J, Cernvall M, Arnberg FK. Efficacy, Benefits, and Harms of a Self-management App in a Swedish Trauma-Exposed Community Sample (PTSD Coach): Randomized Controlled Trial. J Med Internet Res. 2022 Mar 30;24(3):e31419. doi: 10.2196/31419. PMID 35353052